CLINICAL TRIAL: NCT06848777
Title: The Effect of Mobilising Patients Using Nature Sounds on Anxiety, Pain and Stress Levels of Patients After Laparoscopic Cholecystectomy Surgery
Brief Title: The Effect of Mobilising Patients Using Nature Sounds on Anxiety, Pain and Stress Levels
Acronym: After Laparosc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sc129898scy
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Pain; Stress; Laparoscopic Colecctomy; Mobilization; Nature Sound
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To ensure double blinding in this study, patients' anxiety and pain levels were assessed by asking patients questions and having them mark their responses on paper under the supervision of the nurse researcher, while the obtained anxiety and pain scores and the stress levels measured using a smartwatch were recorded on the forms by the independent nurse researcher. The results of the study findings were analyzed by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The standard care protocol of the service will be applied to the patients in the control group. The patients will be mobilized.(
- Intervention Group (Experimental): Patients in this group will be mobilized and will be played nature-based sounds through headphones.
  Interventions: Behavioral: Intervention group:

INTERVENTIONS:
Behavioral: Intervention group: — After a 50-meter walk while listening to the sounds of nature, the patient will walk 50 meters again to his/her room and then to his/her bed, where he/she will be seated. Then, the researcher nurse will remove the headphones from the patient's ears and ensure that the patient rests in a comfortable position.
  Arms: Intervention Group

SUMMARY:
The Effect of Mobilization Using Nature Sounds on Patients' Anxiety, Pain and Stress Levels

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are willing to participate in the study,
* Patients undergoing their first laparoscopic surgery due to gallbladder stones,
* Patients scheduled for elective surgical procedures,
* Patients with no hearing impairment,
* Patients with no vision impairment,
* Mentally stable individuals,
* Individuals who are open to communication and cooperation,
* Patients aged 18 years and older will be included in the study.

Exclusion Criteria:

* Individuals with mental health issues,
* Individuals who are unwilling to participate,
* Patients with hearing impairment,
* Patients undergoing their second surgery (recurrent) due to gallbladder stones,
* Patients using hearing aids,
* Individuals who are uncooperative or unwilling to communicate,
* Patients who require emergency surgery will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Anxiety | Before mobilization 5 minutes and after mobilization 10 minutes
  Anxiety level will be measured withVirtual Analog Scale-Anxiety (The lowest score is set as 0, and the highest score is set as 10.)
Stress | before mobilization 5 minutes and after mobilization 10 minutes
  with smart watch
Pain level | before mobilization 5 minutes and after mobilization 10 minutes
  Pain level will be measured with Virtual Analog Scale (The lowest score is set as 0, and the highest score is set as 10.)

CONTACTS AND LOCATIONS:
Locations (1):
- Kumluca State Hospital, Antalya, Kumluca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided